CLINICAL TRIAL: NCT05376605
Title: ICF-Based Assessment in Lung Transplant Recipients
Brief Title: Assessment of Lung Transplant Recipients Within The Scope of International Classification of Functioning, Disability and Health
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ulaş Ar, MSc, Ankara City Hospital Bilkent
Other Study IDs: E2-21-52
Record Dates: First submitted 2022-05-06; First posted 2022-05-17 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Lung Transplant; Complications; Disability Evaluation
Keywords: International Classification of Functioning, Disability and Health; fatigue; functional capacity
MeSH Terms: conditions — Fatigue | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lung transplant: Patients who have passed at least 3 months after lung transplantation
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment — Evaluations of the patients will be made with scales, questionnaires and physical tests.

SUMMARY:
This study was aimed to evaluate the patients undergoing lung transplantation under the International Classification of Functionality, Disability and Health (ICF) and to examine the relationships between the age at which lung transplant recipients were transplanted and recipients' comorbidity levels and body structure and functions, activity and participation level.

DETAILED DESCRIPTION:
After lung transplantation, many complications related to various reasons are observed in patients in the long term. In this study, the severity of fatigue, limitation of daily living activities, kinesophobia, impaired sleep quality, anxiety and depression level, fragility level, balance and functional capacity in lung transplant recipients; investigators aimed to examine the relationship between the age at which the patient was transplanted and the level of comorbidity. Although there are studies on comorbidities, quality of life, daily living activities and participation level, anxiety and depression level, sleep quality, balance and physical fitness level in lung transplant recipients, kinesiophobia upper extremity functional performance in patients who have undergone lung transplantation surgery, COVID-19 infection There are no studies evaluating the anxiety associated with the disease. No study evaluating body structure functions, activity and participation level based on ICF in lung transplantation has been encountered. In our study, patients with at least 3 months past lung transplantation and without orthopedic and mental problems will be evaluated. It will be made as a single evaluation. The last pulmonary function test results of the patients, comorbidity conditions, fatigue, respiratory quality of life, coronavirus anxiety status, sleep quality, kinesophobia will be evaluated by questionnaires. Lower extremity dynamic balance and mobility will be evaluated with 1 minute sit-to-stand test, timed up and go test. Upper extremity functionality will be evaluated with a 6-minute pegboard and ring test.

ELIGIBILITY:
Inclusion Criteria:

* At least three months have passed since the lung transplantation, without any complications at the last doctor's control
* Clinically stable and, if any, accompanying comorbidities are under control
* Volunteering to participate in research
* Patients who do not have neurological and orthopedic problems that may prevent them from performing functional tests.

Exclusion Criteria:

* Single lung transplant recipient
* Have orthopedic problems
* Patients who cannot cooperate and adapt.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at least 3 months past lung transplantation, who are in stable condition, and who are being followed up by the thoracic surgery clinic of the Ankara city hospital.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Lower extremity exercise capacity assessed by 1 minute sit to stand test (STS) | at least 3 months later post operation
  Number of sit to stands performed by patients in 1 minute
Upper Lower extremity exercise capacity assessed by 6 minutes pegboard and ring test | at least 3 months later post operation
  the number of rings that was moved from the lower pegs to the upper pegs and vice-versa, during a six-minute period
Dyspnea assessed by mMRC dyspnea scale | at least 3 months later post operation
  modified Medical Research Council (mMRC) dyspnea scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing

SECONDARY OUTCOMES:
Sleep quality assessed by Pittsburgh sleep quality index | at least 3 months later post operation
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction
comorbidity level assessed by Charlson comorbidity index | at least 3 months later post operation
  Charlson Comorbidity Index predicts the ten-year mortality for a patient who may have a range of comorbid conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Erdal Yekeler, Professor, Principal Investigator — Ankara City Hospital Bilkent; Ebru Calik-Kutukcu, PhD, Study Director — Hacettepe University Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided